CLINICAL TRIAL: NCT05550207
Title: An Open-Label, Multiple-Dose Evaluation of the Efficacy and Safety of AXS-07 (Meloxicam and Rizatriptan) for the Acute Treatment of Migraine in Adults With a Prior Inadequate Response to an Oral CGRP Inhibitor
Brief Title: Open-Label Study of AXS-07 for the Acute Treatment of Migraine in Adults With a Prior Inadequate Response to an Oral CGRP Inhibitor (EMERGE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXS-07-304
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Migraine
Keywords: Migraine; AXS-07; Meloxicam; Rizatriptan; Oral CGRP inhibitor
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AXS-07 (meloxicam-rizatriptan) (Experimental): Up to 8 weeks
  Interventions: Drug: AXS-07 (meloxicam-rizatriptan)

INTERVENTIONS:
Drug: AXS-07 (meloxicam-rizatriptan) — AXS-07 tablets, taken orally for the acute treatment of migraine

SUMMARY:
This is a multicenter, open-label trial to evaluate the efficacy and safety of AXS-07 in subjects with migraine attacks and prior inadequate response to oral CGRP inhibitors.

DETAILED DESCRIPTION:
Eligible subjects will receive open-label AXS-07 for up to 8 weeks for at-home treatment of their next 4 migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* Has an established diagnosis of migraine with or without aura
* Has experienced an inadequate response to oral CGRP inhibitors for the acute treatment of migraine

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant during the study
* Has previously received any investigational drug or device or investigational therapy within 30 days before Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with headache pain relief | Hour 2 following dose administration
  Absence of headache pain and without the use of rescue medication.
Percentage of subjects with absence of the Most Bothersome Symptom | Hour 2 following dose administration
  Absence of the most bothersome symptom, defined at the onset of migraine.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Clinical Research Site, Colton, California
  - Clinical Research Site, Fullerton, California
  - Clinical Research Site, La Jolla, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Sherman Oaks, California
  - Clinical Research Site, Stamford, Connecticut
  - Clinical Research Site, DeLand, Florida
  - Clinical Research Site, Hallandale, Florida
  - Clinical Research Site, Hollywood, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Ormond Beach, Florida
  - Clinical Research Site, Oviedo, Florida
  - Clinical Research Site, Pensacola, Florida
  - Clinical Research Site, Winter Park, Florida
  - Clinical Research Site, Stockbridge, Georgia
  - Clinical Research Site, Avon, Indiana
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, North Dartmouth, Massachusetts
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Albuquerque, New Mexico
  - Clinical Research Site, The Bronx, New York
  - Clinical Research Site, Williamsville, New York
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Charleston, South Carolina
  - Clinical Research Site, Knoxville, Tennessee
  - Clinical Research Site, Nashville, Tennessee
  - Clinical Research Site, Cypress, Texas
  - Clinical Research Site, Sugar Land, Texas
  - Clinical Research Site, Salt Lake City, Utah
  - Clinical Research Site, Charlottesville, Virginia
  - Clinical Research Site, McLean, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com